CLINICAL TRIAL: NCT01819324
Title: Targeting the Teachable Moment: A Lifestyle Intervention for Breast Cancer Survivors
Brief Title: A Lifestyle Intervention for Breast Cancer Survivors
Acronym: TTMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Park003382HE; 5R21CA152129-02 (NIH)
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: breast cancer survivors; lifestyle intervention; health behaviors
MeSH Terms: conditions — Breast Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Targeting the Teachable Moment (Experimental): Receiving Targeting the Teachable Moment Intervention materials (focusing on health behaviors and issues specific to breast cancer survivors) every other week for 4 months
  Interventions: Behavioral: Targeting the Teachable Moment
- Standardized Lifestyle Management (Active Comparator): Receiving Standardized Lifestyle Management materials (focusing mostly on health behaviors) every other week for 4 months
  Interventions: Behavioral: Standardized Lifestyle Management
- Usual Care (No Intervention): Receiving SLM materials at the end of the 7 months

INTERVENTIONS:
Behavioral: Targeting the Teachable Moment — TTMI material (every other week for 4 months)
  Other Names: TTMI
  Arms: Targeting the Teachable Moment
Behavioral: Standardized Lifestyle Management — SLM material (every other week for 4 months)
  Other Names: SLM
  Arms: Standardized Lifestyle Management

SUMMARY:
1. The purpose of the study is to test the effectiveness of a new mail-based intervention for breast cancer survivors compared with standard lifestyle management and no-treatment.
2. This intervention addresses both lifestyle factors such as dietary and physical activities and psychological issues specific to breast cancer survivors to improve healthy behaviors.

DETAILED DESCRIPTION:
Participants will be assigned randomly to one of three groups: 1) newly developed mail-based intervention (Targeting the Teachable Moment Intervention; TTMI), 2) standard Lifestyle Intervention (SLM), and 3) usual care. Both TTMI and SLM focus on health behaviors, however TTMI additionally addresses psychosocial issues specific to breast cancer survivors.

All participants will complete questionnaires at the time they start the study, the end of the 4 months, and 3 months later for a follow-up.

If participants are assigned to any of the intervention group, they will receive materials every other week for 4 months. If participants are assigned to the usual care group, they will receive the same materials as the standard lifestyle intervention et the end of the 7 months.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosed with breast cancer in the past 1.5 years
* stage 0~2 breast cancer
* no prior adjuvant treatment for another cancer
* Can read and write English
* Are not participating in other health behavior research right now

Exclusion Criteria:

* apparent serious mental disturbance
* male breast cancer survivors

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in eating habits measured by the National Cancer Institute Quick Food Scan | Meaured at baseline, 4 months, and 7 months
  Diet habits (amount of fat and fruit/vegetable uptake) will be assessed at 3 times: at baseline, at the end of the 4 months, and at the end of 7 months.
Changes in physical activity measured by the Paffenbarger physical activity questionnaire | Meaured at baseline, 4 months, and 7 months
  Frequency and amount of time for physical exercise will be measured at 3 times: at baseline, at the end of 4 months, and at the end of 7 months.

SECONDARY OUTCOMES:
Changes in coping strategies measured by the Brief COPE | Measured at baseline, 4 months, and 7 months
  Coping strategies (e.g., problem-focused coping, emotional approach coping) will be assessed at 3 times: at baseline, at the end of the 4 months, and at the end of 7 months.
Changes in Self-efficacy measured by the General Self-Efficacy Scale | Measured at baseline, 4 months, and 7 months
  A general sense of perceived self-efficacy will be measured at 3 times: at the baseline, at the end of 4 months, and at the end of 7 months
Changes in social support measured by the Interpersonal Support Evaluation List (ISEL) | Measured at baseline, 4 months, and 7 months
  Social support will be measured at 3 times: at baseline, at the end of 4 months, and at the end of 7 months
Changes in life meaning measured by the Meaning in Life Questionnaire (MLQ) | Measured at baseline, 4 months, and 7 months
  Presence of Meaning and Search for Meaning will be measured at 3 times: at baseline, at the end of 4 months, and at the end of 7 months.

OTHER OUTCOMES:
Feedback of each module | up to 4 months
  usefulness of each module (e.g., whether each intervention is helpful or not) will be assessed at each mailing (for eight times) for 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L. Park, Ph.D, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States